CLINICAL TRIAL: NCT03671304
Title: Mobile Intervention - Physical Activity in Cancer Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was prematurely discontinued, the application utilized with the fitbit is no longer being supported.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Simmons Cancer Center (Other)
Responsible Party: Principal Investigator, Muhammad Beg, ASSOC PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU 072018-088
Record Dates: First submitted 2018-09-07; First posted 2018-09-14 (Actual); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Carcinoma, Renal Cell
Keywords: renal call carcinoma; exercise; physical activity; mobile intervention; just-in-time adaptive intervention; affective framing; intention planning
MeSH Terms: conditions — Carcinoma, Renal Cell; Motor Activity

STUDY DESIGN:
Intervention Model Description: This project will enroll 50 participants receiving treatment for RCC in an eight-week study. Using a microrandomized design, participants will receive affective framing messages and intention planning prompts on a randomized schedule, such that participants will receive each message type on 50% of days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Just-in-time Adaptive Intervention (Experimental): Participants will receive a Fitbit Versa and instructions on its use. The study design is not a traditional randomized controlled trial in which participants are randomized to either the intervention or control group. Instead the study utilizes a microrandomized design. This is a within-subjects design in which participants will receive affective framing messages and intention planning prompts on a randomized schedule, such that participants will receive each message type on 50% of days.
  Interventions: Device: Fitbit Versa

INTERVENTIONS:
Device: Fitbit Versa — Participants will receive a Fitbit Versa and instructions on its use. Participants will be asked to wear the device for eight weeks, removing it only for charging and when engaging in activities in which the device could be submerged in water (bathing, swimming, etc.).
  At enrollment, participants will indicate a preferred time to receive affective framing messages and EMA prompts (morning), and intention planning prompts (evenings). Participants will receive affective framing messages and intention planning prompts on a randomized schedule, such that participants will receive each message type on 50% of days.

SUMMARY:
Aim 1. Determine the feasibility and acceptability of the proposed mobile technology intervention to increase physical activity patients receiving treatment for renal cell carcinoma.

Aim 2. Evaluate the effect of the proposed intervention components (affective framing, intention planning, and goal-setting) on changes in physical activity.

DETAILED DESCRIPTION:
Recent analyses have indicated that physical activity reduces mortality risk among patients with RCC.1. Physical activity also provides additional benefits for patients undergoing treatment for cancer such as improved quality of life and sleep, and reduced treatment-related fatigue. However, individuals receiving treatment for renal cell carcinoma (RCC) often fail to engage in sufficient physical activity. Many cancer survivors experience a decrease in their physical activity after diagnosis2 and the majority of RCC survivors do not meet the recommended guidelines for physical activity.3 Traditional physical activity interventions require significant resources and present substantial barriers for participants (travel, time commitments, etc.). In contrast, mobile technologies enable delivery of interventions with significantly fewer resources. These technologies also facilitate the delivery of just-in-time adaptive interventions (JITAIs) in which intervention support is provided at only at times when an opportunity for positive changes exists.4 The purpose of this support the development of a JITAI in RCC patients. Evaluation of the acceptability and efficacy of three intervention strategies (affective framing, intention planning, goal-setting, and savoring) will determine their inclusion in the JITAI.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 years or older
2. Diagnosed with RCC
3. < 150 minutes of weekly moderate-to-vigorous physical activity
4. Own a smartphone (required for syncing the Fitbit device).

Exclusion Criteria:

1. Medical condition contraindicating exercise participation
2. Cognitively unable to give informed consent.
3. Unable to read and communicate in English

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Rethorst, BS, Principal Investigator — UT Southwestern
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Just-in-time Adaptive Intervention: Participants will receive a Fitbit Versa and instructions on its use. The study design is not a traditional randomized controlled trial in which participants are randomized to either the intervention or control group. Instead the study utilizes a microrandomized design. This is a within-subjects design in which participants will receive affective framing messages and intention planning prompts on a randomized schedule, such that participants will receive each message type on 50% of days.
  Fitbit Versa: Participants will receive a Fitbit Versa and instructions on its use. Participants will be asked to wear the device for eight weeks, removing it only for charging and when engaging in activities in which the device could be submerged in water (bathing, swimming, etc.).
  At enrollment, participants will indicate a preferred time to receive affective framing messages and EMA prompts (morning), and intention planning prompts (evenings). Participants will receive affective framing messages and intention planning prompts on a randomized schedule, such that participants will receive each message type on 50% of days.
Period: Overall Study
Arm/Group | Just-in-time Adaptive Intervention
Started | 8
Completed | 1
Not Completed | 7
Not completed — study terminated | 7

BASELINE CHARACTERISTICS:
Arm/Group | Just-in-time Adaptive Intervention
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 65 [41 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity (Daily Step Count)
Description: Physical Activity (daily step count) will be measured with the Fitbit.
Time Frame: 8 weeks
Population: Collected data was not considered valid to be analyzed as the application utilized with the fitbit was no longer supported and the study did not complete and was terminated.
Arm/Group | Just-in-time Adaptive Intervention
Number analyzed (Participants) | 0

2. Secondary Outcome: Fitbit Wear Compliance
Description: Assessment of participant compliance with the intervention (days wearing the Fitbit) to determine feasibility for future trials.
Time Frame: 8 weeks
Population: as for outcome 1
Arm/Group | Just-in-time Adaptive Intervention
Number analyzed (Participants) | 0

3. Secondary Outcome: Fitbit Response Compliance
Description: Assessment of participant compliance with the intervention (response rate to intervention prompts) to determine feasibility for future trials.
Time Frame: 8 weeks
Population: as for outcome 1
Arm/Group | Just-in-time Adaptive Intervention
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Adverse events were collected only for approx. 8 weeks because the application utilized with the fitbit was no longer supported and the study did not complete and was terminated.
Arm/Group | Just-in-time Adaptive Intervention
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT03671304/Prot_SAP_000.pdf